CLINICAL TRIAL: NCT04543292
Title: Clinical Evaluation of Polytetrafluoroethylene (PTFE, MATFILL) for the Sealing of Prosthetic Chimneys.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Eduardo Anitua (Other)
Collaborators: BTI Biotechnology Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BTI_01_EP/20/MATFILL; Exp. 812/20/EC (Other: AEMPS)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2020-09

CONDITIONS: Edentulous Alveolar Ridge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MATFILL (Experimental): Prosthetic chimney filling with MATFILL prior to other sealing materials to protect the screww head.
  Interventions: Device: MATFILL (PTFE)

INTERVENTIONS:
Device: MATFILL (PTFE) — Filling of the prosthetic chimney with the compressed material

SUMMARY:
Dental implant supported screwed prosthetic rehabilitations are associated to several advantages, as a minimal occlusal spaced and easier hygiene and maintenance. In this sense, screwed rehabilitations have been associated with lower frequency of biological and technical complications. Nevertheless, the screwing process results in the formation of a prosthetic chimney that requieres an appropriate sealing protocol. This protocol needs to include a material for the protection of the screw head. Nowadays, there is a lack of materials for this intended use with marketing authorisation. Several materials have been tested in the bibliography including PTFE, although there are not high quality studies. In this context, this clinical investigation aims to evaluate the efficacy and safety os a PTFE-based product (MAFILL) for the sealing of prosthetic chimneys and the protection of the screw head.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Clinical need for the placement of a implant-supported dental prosthesis
* Clinical need for the filling of the prosthetic chimney
* Signing informed consent

Exclusion Criteria:

* Inability of follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Integrity of screw head | 6 weeks
  Integrity of the screw head observed in photographs
Integrity of screw head | 6 weeks
  Retightening after screw after unscrew

SECONDARY OUTCOMES:
Occurrence of prosthetic complications | 6 weeks
  Occurrence of prosthetic complications during follow-up
Occurrence of biological complications | 6 weeks
  Occurrence of biological complications

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Anitua, MD, DDS, PhD, Principal Investigator — Eduardo Anitua Private Clinic
Locations (1):
- Eduardo Anitua Private Clinic, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No